CLINICAL TRIAL: NCT07263334
Title: The Effect of Text Neck Syndrome on the Muscle and Bone Architecture of the Cervical Region
Brief Title: Does Mental Fatigue Caused by Social Media Use Affect Biomechanical Properties of Muscles in Young Male Athletes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Asoc. Prof, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-110
Record Dates: First submitted 2025-03-22; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Mental Fatigue; Socail Media Usage; Cervical Range of Motion
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Some of the researchers (O.B.T., B.A., M.B.U.) performed all assessments. To avoid any bias, group information was kept confidential,and statistical analyses were performed by another researcher (A.K., B.Ç., A.G.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Design (Experimental): The study was conducted as a single-blind experimental study. Since it was thought that mental functions might be affected, all the procedures to be applied were explained to the participants, and written informed consent was obtained, but the purpose and hypotheses were not explained. After the final assessment of the participants was completed, the purpose and hypotheses of this study were explained. The study was conducted between June 2024 and February 2025.
  Interventions: Other: Metal Fatigue Protocols

INTERVENTIONS:
Other: Metal Fatigue Protocols — Metal Fatigue Protocols Participants used Instagram® for 30 minutes by browsing their personal feed with one-handed tapping and swiping gestures. They were allowed to scroll and like posts but were restricted from viewing stories or reels and from sharing any content.

SUMMARY:
The aim of this study is to examine the effect of mental fatigue (MF) induced by 30 minutes of social media use on neck kinematics and neck muscle biomechanical properties in young male athletes. Twenty-five participants are enrolled in a single-blind cross-sectional design. Baseline and post-MF assessments include cervical range of motion measured with a CROM device, forward head posture evaluated using craniovertebral angle analysis, and muscle tone, stiffness, and elasticity measured with MyotonPRO. MF is induced through 30 minutes of Instagram® use on a smartphone and quantified with a 100-mm Visual Analogue Scale (VAS). No results or conclusions are provided in this section.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of mental fatigue (MF) induced by 30 minutes of social media use on neck kinematics and the biomechanical properties of the neck muscles [upper trapezius, sternocleidomastoid (SCM), semispinalis (SS), and splenius capitis (SC)] in young male athletes. Twenty-five young male athletes are enrolled in a single-blind cross-sectional study. Participants undergo assessments at baseline and again following MF induction. These assessments include cervical range of motion (CROM) measured with a validated CROM device, forward head posture (FHP) evaluated via craniovertebral angle (CVA) photometric analysis, and muscle biomechanical properties (tone, stiffness, elasticity) measured using the MyotonPRO device. Mental fatigue is induced through 30 minutes of Instagram use on a smartphone. MF severity is assessed using a 100-mm Visual Analogue Scale (VAS). No results or conclusions are reported in this section.

ELIGIBILITY:
Inclusion Criteria:

* Amateur athletes aged 18-35
* using social media via a smartphone
* actively participating in competitions

Exclusion Criteria:

* having a surgical operation or trauma related to the neck region, having any pathology in the neck region (neck cyst, tumours, haematoma, etc.), having a history of traumatic injury in the neck region, and having neurological and rheumatic diseases.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Range of Motion of the Neck | Baseline
  The normal joint motion of the cervical region was evaluated with the Cervical Range of Motion (CROM-Perfomance Attainment Associates, St. Paul, MN, 55117, United States) device, which has clinical validity and reliability. The flexion, extension, right and left lateral flexion and rotation angles of the cervical region were measured three times and averaged with the CROM device.
Forward Head Posture | Baseline
  The craniovertebral angle (CVA) was measured using a photometric method with the participants in a standing position. Prior to imaging, the C7 process and tragus were marked. A camera was placed 1.5 m from the lateral surface of the body at the level of the acromial process.
Biomechanical Properties of Muscles | Baseline
  The biomechanical properties of cervical muscles were assessed using the MyotonPRO, which quantifies tissue oscillations following a brief mechanical impulse to determine tone, stiffness, and elasticity. This method provides reliable interrater and intrarater measurements for cervical musculature when applied perpendicularly in a standardized supine position, as demonstrated in previous research. For each muscle, three consecutive measurements were recorded following established protocols for the sternocleidomastoid and upper trapezius.The MyotonPro enables the assessment of various parameters, including the state of resting muscle tone (F), defined as the suppressed EMG signal, and dynamic stiffness (S). The basis of stiffness assessment using myotonometry is the theory of free oscillations, arising from the natural oscillations of tissues in response to brief mechanical exposure of the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciencies, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No